CLINICAL TRIAL: NCT06551805
Title: Clinical Research Protocol of Ferumoxytol for Magnetic Resonance Enhancement Imaging in Patients With Atherosclerosis.
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-178-05
Record Dates: First submitted 2023-06-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — ferumoxides

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Safety assessment and the diagnostic value of Ferumoxytol.: Drug Name: Ferumoxytol Dosage Form: Injection Dosage: 3 mg/kg Administration Frequency: Single intravenous injection
  Interventions: Drug: Safety assessment of Ferumoxytol.; Drug: Assessment of the diagnostic value of Ferumoxytol for MR angiography.

INTERVENTIONS:
Drug: Safety assessment of Ferumoxytol. — Observe the injection site for skin invagination, rash, or urticaria during injection. Patients and their relatives were asked about any subjective adverse events before, during, and after drug injection, and all adverse events were recorded on the case report forms, and adverse events were scored according to the Common Terminology Criteria for Adverse Events (CTCAE) from Grade 1 "mild" to Grade 5 "death", Observe the vital signs of patients. Patients undergoing MRI underwent electrocardiogram (ECG) monitoring before and within 60 minutes after ferumoxytol administration, specifically including: biochemical panel, iron metabolism, liver and kidney function, cytokines, blood routine, urine routine, 24-hour urine volume, glycosylated hemoglobin and so on. All patients received a total of 3 blood and urine collections at 7 days before injection, 48 hours after injection, 1month to 3months after injection.
  Other Names: Superparamagnetic iron oxide
Drug: Assessment of the diagnostic value of Ferumoxytol for MR angiography. — steady-state, high-spatial-resolution, three-dimensional fast low-angle shot acquisition technique, T2W-MDIR imaging, polysaccharide superparamagnetic iron oxide injection enhanced T1W and T2W, T2* mapping, and Steady state free precession sequence, T2 weighted black blood sequence, T2 preparation single shot steady state free precession sequence, T2* weighted multi-echo/gradient echo sequence, polysaccharide superparamagnetic iron oxide injection enhanced imaging, Breath-triggered Transverse 3D Balance-Vortex Field Echo (b-TFE) Magnetic Resonance Angiography, iMSDE-SPGR Sequence, 4D Flow MRI. the MRI anxiety questionnaire.
  Other Names: Superparamagnetic iron oxide

SUMMARY:
We are preparing to initiate a clinical trial involving Ferumoxytol for magnetic resonance-enhanced imaging in patients with atherosclerosis. The aim of this study is to assess the safety and effectiveness of Ferumoxytol for magnetic resonance angiography in patients with atherosclerosis.

DETAILED DESCRIPTION:
In this study, the safety of Ferumoxytol as an MR imaging contrast agent will be assessed by monitoring vital signs and laboratory parameters such as complete blood count, urinalysis, and liver and kidney function tests before and after administration of Ferumoxytol. Following the injection, all patients will undergo two MRI scans at different time intervals, ranging from 0 to 15 hours and from 24 to 48 hours. Within one week prior to the injection, patients will undergo standard laboratory tests as part of their routine clinical assessment, and the pre-administration lab results will be documented.

This study will prospectively enroll patients with atherosclerosis, and Ferumoxytol-enhanced MRA imaging will be performed on all patients to investigate the diagnostic utility of Ferumoxytol as an MR imaging contrast agent.

ELIGIBILITY:
Inclusion criteria: Patients aged 18 years and older with atherosclerosis.

Exclusion criteria:

Individuals with a history of allergy or hypersensitivity to iron or dextran. Patients currently receiving oral or intravenous iron therapy. Patients with hemosiderosis or hemochromatosis. Patients with a history of allergic reactions to intravenous iron products or any iron overload-related conditions.

Individuals who are unable to undergo magnetic resonance imaging (MRI) due to psychological reasons (such as claustrophobia) or physical reasons (such as the presence of non-compatible metallic objects in the body).

Patients with end-stage diseases or life expectancy less than 1 year. Pregnant women. Any other individuals deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. CKD patients aged ≥18 years.
  2. Presence of atherosclerosis in the head and neck vessels and/or coronary arteries and/or renal arteries, as indicated by other evidence.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Ferumoxytol demonstrates a favorable safety profile in human subjects. | 2023.10-2026.12
  safe
Ferumoxytol exhibits diagnostic efficacy for MR angiography. | 2023.10-2026.12
  diagnostic efficacy

OTHER OUTCOMES:
lower limb artery Image Acquisition | All patients underwent MRI after injection of polysaccharide superparamagnetic iron oxide injection.
  atherosclerosis
Adverse Events | Before, during, after injection
  no adverse events
Vital signs | Obtained before injection, 15, 30, 45, 60 minutes after injection and before and after the second MR scan.
  safety

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fraum TJ, Ludwig DR, Bashir MR, Fowler KJ. Gadolinium-based contrast agents: A comprehensive risk assessment. J Magn Reson Imaging. 2017 Aug;46(2):338-353. doi: 10.1002/jmri.25625. Epub 2017 Jan 13. PMID 28083913
- [Background] McDonald RJ, Levine D, Weinreb J, Kanal E, Davenport MS, Ellis JH, Jacobs PM, Lenkinski RE, Maravilla KR, Prince MR, Rowley HA, Tweedle MF, Kressel HY. Gadolinium Retention: A Research Roadmap from the 2018 NIH/ACR/RSNA Workshop on Gadolinium Chelates. Radiology. 2018 Nov;289(2):517-534. doi: 10.1148/radiol.2018181151. Epub 2018 Sep 11. PMID 30204075
- [Background] Blomqvist L, Nordberg GF, Nurchi VM, Aaseth JO. Gadolinium in Medical Imaging-Usefulness, Toxic Reactions and Possible Countermeasures-A Review. Biomolecules. 2022 May 24;12(6):742. doi: 10.3390/biom12060742. PMID 35740867
- [Background] Idee JM, Port M, Robic C, Medina C, Sabatou M, Corot C. Role of thermodynamic and kinetic parameters in gadolinium chelate stability. J Magn Reson Imaging. 2009 Dec;30(6):1249-58. doi: 10.1002/jmri.21967. PMID 19938037
- [Background] Kanda T, Ishii K, Kawaguchi H, Kitajima K, Takenaka D. High signal intensity in the dentate nucleus and globus pallidus on unenhanced T1-weighted MR images: relationship with increasing cumulative dose of a gadolinium-based contrast material. Radiology. 2014 Mar;270(3):834-41. doi: 10.1148/radiol.13131669. Epub 2013 Dec 7. PMID 24475844
- [Background] Roberts DR, Holden KR. Progressive increase of T1 signal intensity in the dentate nucleus and globus pallidus on unenhanced T1-weighted MR images in the pediatric brain exposed to multiple doses of gadolinium contrast. Brain Dev. 2016 Mar;38(3):331-6. doi: 10.1016/j.braindev.2015.08.009. Epub 2015 Sep 4. PMID 26345358
- [Background] Miller JH, Hu HH, Pokorney A, Cornejo P, Towbin R. MRI Brain Signal Intensity Changes of a Child During the Course of 35 Gadolinium Contrast Examinations. Pediatrics. 2015 Dec;136(6):e1637-40. doi: 10.1542/peds.2015-2222. Epub 2015 Nov 16. PMID 26574593
- [Background] Muehe AM, Feng D, von Eyben R, Luna-Fineman S, Link MP, Muthig T, Huddleston AE, Neuwelt EA, Daldrup-Link HE. Safety Report of Ferumoxytol for Magnetic Resonance Imaging in Children and Young Adults. Invest Radiol. 2016 Apr;51(4):221-227. doi: 10.1097/RLI.0000000000000230. PMID 26656202
- [Background] Spinowitz BS, Kausz AT, Baptista J, Noble SD, Sothinathan R, Bernardo MV, Brenner L, Pereira BJ. Ferumoxytol for treating iron deficiency anemia in CKD. J Am Soc Nephrol. 2008 Aug;19(8):1599-605. doi: 10.1681/ASN.2007101156. Epub 2008 Jun 4. PMID 18525001
- [Background] Hope MD, Hope TA, Zhu C, Faraji F, Haraldsson H, Ordovas KG, Saloner D. Vascular Imaging With Ferumoxytol as a Contrast Agent. AJR Am J Roentgenol. 2015 Sep;205(3):W366-73. doi: 10.2214/AJR.15.14534. Epub 2015 Jun 23. PMID 26102308
- [Background] Kooi ME, Cappendijk VC, Cleutjens KB, Kessels AG, Kitslaar PJ, Borgers M, Frederik PM, Daemen MJ, van Engelshoven JM. Accumulation of ultrasmall superparamagnetic particles of iron oxide in human atherosclerotic plaques can be detected by in vivo magnetic resonance imaging. Circulation. 2003 May 20;107(19):2453-8. doi: 10.1161/01.CIR.0000068315.98705.CC. Epub 2003 Apr 28. PMID 12719280
- [Background] Bashir MR, Bhatti L, Marin D, Nelson RC. Emerging applications for ferumoxytol as a contrast agent in MRI. J Magn Reson Imaging. 2015 Apr;41(4):884-98. doi: 10.1002/jmri.24691. Epub 2014 Jun 30. PMID 24974785
- [Background] Stephen ZR, Kievit FM, Zhang M. Magnetite Nanoparticles for Medical MR Imaging. Mater Today (Kidlington). 2011 Jul;14(7-8):330-338. doi: 10.1016/S1369-7021(11)70163-8. PMID 22389583
- [Background] Jeon M, Halbert MV, Stephen ZR, Zhang M. Iron Oxide Nanoparticles as T1 Contrast Agents for Magnetic Resonance Imaging: Fundamentals, Challenges, Applications, and Prospectives. Adv Mater. 2021 Jun;33(23):e1906539. doi: 10.1002/adma.201906539. Epub 2020 Jun 4. PMID 32495404
- [Background] Blockley NP, Jiang L, Gardener AG, Ludman CN, Francis ST, Gowland PA. Field strength dependence of R1 and R2* relaxivities of human whole blood to ProHance, Vasovist, and deoxyhemoglobin. Magn Reson Med. 2008 Dec;60(6):1313-20. doi: 10.1002/mrm.21792. PMID 19030165
- [Background] Nayak AB, Luhar A, Hanudel M, Gales B, Hall TR, Finn JP, Salusky IB, Zaritsky J. High-resolution, whole-body vascular imaging with ferumoxytol as an alternative to gadolinium agents in a pediatric chronic kidney disease cohort. Pediatr Nephrol. 2015 Mar;30(3):515-21. doi: 10.1007/s00467-014-2953-x. Epub 2014 Sep 12. PMID 25212105
- [Background] Walker JP, Nosova E, Sigovan M, Rapp J, Grenon MS, Owens CD, Gasper WJ, Saloner DA. Ferumoxytol-enhanced magnetic resonance angiography is a feasible method for the clinical evaluation of lower extremity arterial disease. Ann Vasc Surg. 2015 Jan;29(1):63-8. doi: 10.1016/j.avsg.2014.09.003. Epub 2014 Sep 28. PMID 25269682
- [Background] Ruangwattanapaisarn N, Hsiao A, Vasanawala SS. Ferumoxytol as an off-label contrast agent in body 3T MR angiography: a pilot study in children. Pediatr Radiol. 2015 Jun;45(6):831-9. doi: 10.1007/s00247-014-3226-3. Epub 2014 Nov 27. PMID 25427433
- [Background] Li W, Tutton S, Vu AT, Pierchala L, Li BS, Lewis JM, Prasad PV, Edelman RR. First-pass contrast-enhanced magnetic resonance angiography in humans using ferumoxytol, a novel ultrasmall superparamagnetic iron oxide (USPIO)-based blood pool agent. J Magn Reson Imaging. 2005 Jan;21(1):46-52. doi: 10.1002/jmri.20235. PMID 15611942
- [Background] Wilson S, Culp WTN, Wisner ER, Cissell DD, Finn JP, Zwingenberger AL. Ferumoxytol-enhanced magnetic resonance angiography provides comparable vascular conspicuity to CT angiography in dogs with intrahepatic portosystemic shunts. Vet Radiol Ultrasound. 2021 Jul;62(4):463-470. doi: 10.1111/vru.12963. Epub 2021 Feb 26. PMID 33634935
- [Background] Stoumpos S, Tan A, Hall Barrientos P, Stevenson K, Thomson PC, Kasthuri R, Radjenovic A, Kingsmore DB, Roditi G, Mark PB. Ferumoxytol MR Angiography versus Duplex US for Vascular Mapping before Arteriovenous Fistula Surgery for Hemodialysis. Radiology. 2020 Oct;297(1):214-222. doi: 10.1148/radiol.2020200069. Epub 2020 Jul 21. PMID 32692301
- [Background] Yilmaz A, Dengler MA, van der Kuip H, Yildiz H, Rosch S, Klumpp S, Klingel K, Kandolf R, Helluy X, Hiller KH, Jakob PM, Sechtem U. Imaging of myocardial infarction using ultrasmall superparamagnetic iron oxide nanoparticles: a human study using a multi-parametric cardiovascular magnetic resonance imaging approach. Eur Heart J. 2013 Feb;34(6):462-75. doi: 10.1093/eurheartj/ehs366. Epub 2012 Oct 26. PMID 23103659
- [Background] Mukundan S, Steigner ML, Hsiao LL, Malek SK, Tullius SG, Chin MS, Siedlecki AM. Ferumoxytol-Enhanced Magnetic Resonance Imaging in Late-Stage CKD. Am J Kidney Dis. 2016 Jun;67(6):984-8. doi: 10.1053/j.ajkd.2015.12.017. Epub 2016 Jan 16. PMID 26786296